CLINICAL TRIAL: NCT04124185
Title: Phenotyping and Genotyping Patients With Achromatopsia in Preparation for Gene Therapy Trials
Brief Title: Natural History Study for Achromatopsia
Status: Completed | Type: Observational
Sponsor: MeiraGTx UK II Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MGT008
Record Dates: First submitted 2019-09-10; First posted 2019-10-11 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Achromatopsia
Keywords: Achromatopsia; CNGB3; CNGA3
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples for genetic screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Achromatopsia
  Interventions: Diagnostic Test: Ocular assessments

INTERVENTIONS:
Diagnostic Test: Ocular assessments — Complete ocular examination, Axial length and corneal curvature, Optical Coherence Tomography, Visual acuity, Contrast sensitivity

SUMMARY:
In preparation for human clinical trials we intend to undertake a detailed phenotypic study to help to identify patients who may be suitable for therapeutic intervention. In addition, with the recent availability of advanced imaging modalities, further detailed phenotypic investigations will also be valuable in helping to probe the relationship between structure and function and may shed light on disease mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with molecularly proven Achromatopsia or a typical clinical Achromatopsia phenotype with genetic screening pending.
* Minimum subject age of 3 years.
* Able to give consent/parent or guardian able to give consent.

Exclusion Criteria:

* Patients unable or unwilling to undertake consent or clinical testing.
* Patients unwilling to donate a blood sample in order to establish the genetic cause of their condition.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Achromatopsia
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Complete ocular examination | 5 years
Axial length | 5 years
Corneal curvature | 5 years
Optical Coherence Tomography | 5 years
Visual acuity | 5 years
Contrast sensitivity | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided